CLINICAL TRIAL: NCT02302573
Title: Placenta Accreta : Contrast-enhanced Ultrasound Analysis in High Risk Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHRI08-FP : Placenta Accreta
Record Dates: First submitted 2014-11-14; First posted 2014-11-27 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2016-12

CONDITIONS: Placenta Accreta
Keywords: placenta accreta; contrast-enhanced unltrasound; pregnancy; MRI; sonovue
MeSH Terms: conditions — Placenta Accreta | interventions — contrast agent BR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- placenta accreta (Experimental): contast-enhanced ultrasound with sonovue
  Interventions: Drug: contast-enhanced ultrasound with sonovue

INTERVENTIONS:
Drug: contast-enhanced ultrasound with sonovue — contast-enhanced ultrasound with sonovue
  Other Names: Sonovue® (Bracco, Milan, Italie)

SUMMARY:
Abnormally invasive placenta (AIP) is defined as an abnormal placental attachment of a part or the entire chorionic plate with penetration of chorionic villi in the myometrium and absence of the decidua basalis. This anomaly is associated with significant maternal morbidity and mortality as it may result in severe haemorrhage during the post-partum. It has been demonstrated that prenatal diagnosis of AIP is essential to reduce maternal morbidity. In a recent study of Chantraine F. et al. prenatal diagnosis of AIP leads to better outcomes, due to fewer emergency operations and less mass transfusions. Currently, the diagnosis of AIP is based on a combination of conventional B-mode ultrasound and MRI. However, prenatal diagnosis of AIP remains challenging and recent reports demonstrated it is achieved in only thirds of cases.

Contrast enhanced ultrasound (CEUS) is a non-invasive technique based on the detection by ultrasound (US) of gas-filled microbubbles used as perfusion tracers. Intravascular rheological properties of these bubbles are similar to those of red blood cells and they remain entirely within the intravascular space. Previous studies have demonstrated that microbubbles do not transfer into fetal circulation. CEUS has been used for years in many US imaging applications (e.g. liver, kidneys and breast). In obstetrics, despite not yet approved for clinical use, CEUS offers the opportunity to analyze anatomical placental landmarks, improving the contrast between placenta and myometrium. In addition, quantification parameters related to the contrast enhancement have been proposed as objective indicators to estimate blood perfusion rates in the placental intervillous space.

The main objective of this study is to provide pre-clinical evaluation of CEUS for the diagnosis of AIP and to try to determine if AIP are characterised by differences in intervillous blood rheological properties. Conventional CEUS parameters will be: rise time, peak enhancement, wash-in rate, mean transit time and wash-in area under the curve.

As this study is a pre-clinical evaluation, sample size calculation remains subjective and imprecise. For this reason, a sample size of 100 pregnant women to be included in this prospective study has been decided.

The potential impact of this study will be to propose a more reliable tool with both improved sensibility and specificity compared to the combination US/MRI and therefore to reduce the maternal worldwide burden of AIP.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patient having any of the following two conditions:

  * Scar uterus (previous cesarean) with placenta previa partly or wholly on the uterine scar
  * Placenta praevia and patient aged over 35 years
* Term > 34 weeks of amenorrhea
* More than 18 years old
* Inform consent form signed
* affiliated to medical insurrance

Exclusion Criteria:

* Inability to understand information
* Contraindications to the contrast medium Sonovue:
* Hypersensitivity to hexafluorinated sulphur or any other components of Sonovue

  * Recent acute coronary syndrome (within 6 months before the intervention)
  * Unstable ischemic heart disease (myocardial infarction being formed or evolving, typical angina of rest in the previous month)
  * Significant worsening of cardiac symptoms between the pre anaesthesia consultation and intervention
  * Recent intervention (less than 6 months) on coronary arteries or other factor suggesting clinical instability (changes in ECG, changes in clinical or biological parameters)
  * Acute heart failure or heart failure stage III or IV
  * Severe arrhythmias
  * Right-left shunt
  * Acute endocarditis
  * Valve prothesis
  * Severe pulmonary hypertension (pulmonary artery pressure > 90mmHg)
  * Systemic hypertension uncontrolled
  * Respiratory distress syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-05; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Conventional contrast enhanced ultrasound parameters for diagnosing placenta accreta | up to 9 months after consent

SECONDARY OUTCOMES:
depth of infiltration placenta measured by CEUS | up to 9 months after consent

CONTACTS AND LOCATIONS:
Overall Officials: Franck Perrotin, MD, Principal Investigator — University Hospital of Tours
Locations (2):
- France (2):
  - CHU La Millétrie, Poitiers
  - University Hospital of Tours, Tours

REFERENCES:
- [Result] Denis de Senneville B, Novell A, Arthuis C, Mendes V, Dujardin PA, Patat F, Bouakaz A, Escoffre JM, Perrotin F. Development of a Fluid Dynamic Model for Quantitative Contrast-Enhanced Ultrasound Imaging. IEEE Trans Med Imaging. 2018 Feb;37(2):372-383. doi: 10.1109/TMI.2017.2743099. Epub 2017 Aug 29. PMID 28858788